CLINICAL TRIAL: NCT00542945
Title: A DANish Randomized, Controlled, Multicenter Study to Assess the Efficacy of Implantable Cardioverter Defibrillator in Patients With Non-ischemic Systolic Heart Failure on Mortality. The DANISH Study
Brief Title: Danish ICD Study in Patients With Dilated Cardiomyopathy
Acronym: DANISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Study Group (Network)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Danish-ICD-001
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Dilated Cardiomyopathy; Reduced LVEF
Keywords: Heart Failure; ICD; Dilated cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Heart Failure nonischemic ethiology
  Interventions: Device: ICD
- B (Active Comparator)
  Interventions: Other: Optimal medical treatment

INTERVENTIONS:
Device: ICD — Implantation of an ICD
  Arms: A
Other: Optimal medical treatment — ACE-inhibitors or ARB Beta-blocker Optional aldosterone antagonist
  Arms: B

SUMMARY:
The primary objective of this study is to determine the efficacy of ICD therapy compared with control on the endpoint of death from any cause in patients with heart failure of non-ischemic oetiology.

DETAILED DESCRIPTION:
Title: A DANish randomized, controlled, multicenter study to assess the efficacy of Implantable cardioverter defibrillator in patients with non-ischemic Systolic Heart failure on mortality.

Indication: Prevention of mortality in patients at risk of sudden death.

Primary objective: The primary objective of this study is to determine the efficacy of ICD therapy compared with control on the endpoint of death from any cause.

Secondary objective: The secondary objectives of the study are to determine if ICD therapy reduces sudden death.

Study design: Randomized, unblinded, controlled, parallel two group trial.

Primary endpoint: Time to death from any cause.

Sample size: In total, 1000 patients with 500 receiving ICD and 500 patients constituting the control group.

Summary of Subject Eligibility Criteria: Patients with clinical heart failure, left ventricular ejection fraction (LVEF) ≤ 35%, non-ischemic ethiology and NT-proBNP above 200 pg/ml. Patients in NYHA class IV will only be randomised if also fulfilling criteria for a biventricular pacemaker.

Control group: Patients receiving standard therapy for heart failure including ACE-inhibitor/Angiotensin-Receptor-Blocker and Betablocker unless not tolerated. Aldosterone antagonism is optional.

Study Duration: The study comprises a screening period of up to 2 years, followed by a treatment phase of a minimum of 36 months.

Screening and Randomisation: After the signing of informed consent, screening will include medical history, vital signs, physical exam, blood chemistry, haematology, and NT-proBNP. After fulfilling all eligibility criteria, subjects will be randomized 1:1 to receive ICD implantation or continue usual control. Randomisation will be stratified according to treatment with a biventricular pacemaker.

Treatment: After randomisation patients allocated to ICD treatment should receive this as fast as possible and preferably within 2 weeks (latest 4 weeks). The ICD will be programmed with anti-tachycardia pacing and shock therapy.

Assessments: Deaths and hospitalisations for heart failure, stroke or arrhythmias will be recorded throughout the study duration. An Endpoint Classification Committee will adjudicate hospitalizations and deaths for causality.

An independent Data Monitoring Committee will periodically review mortality data throughout the study.

Statistical Considerations: Median lifetime in the control group is expected to be 5 years. A p-value of 5% (2-sided) is required for significance together with a power of at least 80%. With a relative risk reduction of 25% a sample size of 812 patients in total is required. In order to allow for cross-over a sample size of 1000 is planned.

Primary Endpoint Analysis: The principal analysis for the primary endpoint (time to death from any cause) will employ the intent-to-treat principle and use a survival analysis. For each treatment group, Kaplan-Meier curves will be estimated, graphically displayed, and compared using a logrank test. A covariate-adjusted analysis of the primary endpoint using a Cox proportional hazards model will be performed as a supportive analysis. The hazard ratio and its corresponding 95% confidence interval will be estimated. Subjects withdrawing from the study early (other than for withdrawal of consent) will be followed for potential development of the primary endpoint. Subjects completing the study and not experiencing the composite event will be censored.

Secondary Endpoint Analysis: All time-to-event secondary endpoints will be analyzed similarly to the primary endpoint.

Sample Size: Hazard rates have been estimated for the placebo and ICD groups using subjects from a variety of databases (including the Echos database and the publication of Definite). Assuming a 24-month enrollment period and a 36 month follow-up period (resulting in a 5-year study with a minimum treatment period of 3 years and approximately a median survival time of 60 months), a total of 812 subjects will provide a 80% power with a 2-sided significance level of 5% for detecting a reduction in hazard of 25%.

Safety Summary: The subject incidence of adverse events will be tabulated for each group. Adverse events related to ICD implantation will be summarized. During the trial inappropriate shocks will be summarized.

Data Monitoring Committee: An independent Data Monitoring Committee consisting of members with relevant expertise will be assembled prior to study commencement. This committee will periodically review safety data.

Endpoint Classification Committee: An external Endpoint Classification Committee will adjudicate death as sudden or non-sudden throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of screening.
* Documented non-ischemic HF with an LVEF ≤ 35%.
* NYHA class II-III. If patients are planned for an implantation with a biventricular pacemaker NYHA class IV patients will be accepted for the trial.
* Before any study-specific procedure, including assessments for screening, the appropriate written informed consent must be obtained (see section 12.1).
* NT-proBNP above 200 pg/ml (see appendix D).

Exclusion Criteria:

To be eligible for this study, subjects must not meet any of the following criteria:

* Uncorrected congenital heart disease or valve obstruction, obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, untreated hypothyroidism or hyperthyroidism, adrenal insufficiency, active vasculitis due to collagen vascular disease.
* On the urgent waiting list for a heart transplant (UNOS category 1A or 1B, or equivalent). Patients on the non-urgent waiting list for a heart transplant (UNOS category 2 or 7, or equivalent) are eligible for inclusion in the study.
* Recipient of any major organ transplant (eg, lung, liver, heart or kidney).
* Receiving or has received cytotoxic or cytostatic chemotherapy and/or radiation therapy for treatment of a malignancy within 6 month before randomisation or clinical evidence of current malignancy, with the following exceptions: basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, prostate cancer (if stable localized disease, with a life expectancy of > 2.5 years in the opinion of the investigator).
* Known to be human immunodeficiency virus positive with an expected survival of less than 5 years due to HIV.
* Renal failure treated with dialysis.
* Recent (within 3 months) history of alcohol or illicit drug abuse disorder, based on self-report
* Any condition (eg, psychiatric illness) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 5 years

SECONDARY OUTCOMES:
Quality of Life and health economics | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Køber, MD, D.Sci, Study Chair — Department of Cardiology, Rigshospitalet.
Locations (1):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Butt JH, Doi SN, Thune JJ, Nielsen JC, Videbaek L, Yafasova A, Bruun NE, Torp-Pedersen C, Eiskjaer H, Egstrup K, Brandes A, Hassager C, Svendsen JH, Hofsten D, Pehrson S, Kober L. Long-Term Effect of ICDs in Nonischemic Heart Failure With Reduced Ejection Fraction: Extended Follow-Up Analysis of DANISH. J Am Coll Cardiol. 2025 Dec 16;86(24):2402-2414. doi: 10.1016/j.jacc.2025.08.089. Epub 2025 Oct 22. PMID 41123523
- [Derived] Butt JH, Bundgaard JS, Schou M, Yafasova A, Doi SN, Svendsen JH, Hofsten DE, Hassager C, Eiskjaer H, Nielsen JC, Bruun NE, Videbaek L, Brandes A, Thune JJ, Pehrson S, Kober L. Implantable Cardioverter-Defibrillator and Frailty in Non-ischemic Heart Failure With Reduced Ejection Fraction: Extended Follow-Up of the DANISH Trial. Am J Cardiol. 2026 Jan 15;259:163-172. doi: 10.1016/j.amjcard.2025.08.068. Epub 2025 Sep 23. PMID 40998196
- [Derived] Doi SN, Yafasova A, Thune JJ, Nielsen JC, Bruun NE, Videbaek L, Eiskjaer H, Hassager C, Svendsen JH, Hofsten DE, Pehrson S, Kober L, Butt JH. Atrial fibrillation and implantable cardioverter-defibrillator in non-ischaemic heart failure with reduced ejection fraction: insights from the DANISH trial. Europace. 2025 Sep 1;27(9):euaf200. doi: 10.1093/europace/euaf200. PMID 40990042
- [Derived] Butt JH, Thune JJ, Nielsen JC, Haarbo J, Videbaek L, Gustafsson F, Kristensen SL, Bruun NE, Eiskjaer H, Brandes A, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Schou M, Pehrson S, Packer M, McMurray JJV, Kober L. Anthropometric measures and long-term mortality in non-ischaemic heart failure with reduced ejection fraction: Questioning the obesity paradox. Eur J Heart Fail. 2025 Mar;27(3):527-536. doi: 10.1002/ejhf.3424. Epub 2024 Aug 18. PMID 39155576
- [Derived] Karacan MN, Doi SN, Yafasova A, Thune JJ, Nielsen JC, Haarbo J, Bruun NE, Gustafsson F, Eiskjaer H, Hassager C, Svendsen JH, Hofsten DE, Pehrson S, Kober L, Butt JH. New York Heart Association functional class and implantable cardioverter-defibrillator in non-ischaemic heart failure with reduced ejection fraction: Extended follow-up of the DANISH trial. Eur J Heart Fail. 2024 Jun;26(6):1423-1431. doi: 10.1002/ejhf.3239. Epub 2024 May 11. PMID 38733253
- [Derived] Doi SN, Thune JJ, Nielsen JC, Haarbo J, Videbaek L, Yafasova A, Bruun NE, Gustafsson F, Eiskjaer H, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S, Kober L, Butt JH. Estimated Glomerular Filtration Rate and Implantable Cardioverter-Defibrillator in Nonischemic Systolic Heart Failure: Extended Follow-Up of DANISH. J Am Heart Assoc. 2024 Feb 6;13(3):e031977. doi: 10.1161/JAHA.123.031977. Epub 2024 Jan 31. PMID 38293926
- [Derived] Butt JH, Yafasova A, Doi SN, Nielsen JC, Haarbo J, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Hassager C, Svendsen JH, Hofsten DE, Videbaek L, Torp-Pedersen C, Pehrson S, Thune JJ, Kober L. Implantable Cardioverter Defibrillator in Patients With Nonischemic Systolic Heart Failure With and Without Cardiac Resynchronization Therapy: Extended Follow-Up Study of the DANISH Trial. Circulation. 2023 Oct 10;148(15):1179-1181. doi: 10.1161/CIRCULATIONAHA.123.065560. Epub 2023 Oct 9. No abstract available. PMID 37812653
- [Derived] Butt JH, Yafasova A, Elming MB, Dixen U, Nielsen JC, Haarbo J, Videbaek L, Korup E, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Egstrup K, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S, Thune JJ, Kober L. Efficacy of Implantable Cardioverter Defibrillator in Nonischemic Systolic Heart Failure According to Sex: Extended Follow-Up Study of the DANISH Trial. Circ Heart Fail. 2022 Sep;15(9):e009669. doi: 10.1161/CIRCHEARTFAILURE.122.009669. Epub 2022 Aug 9. PMID 35942877
- [Derived] Butt JH, Yafasova A, Elming MB, Dixen U, Nielsen JC, Haarbo J, Videbaek L, Korup E, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Egstrup K, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S, Thune JJ, Kober L. NT-proBNP and ICD in Nonischemic Systolic Heart Failure: Extended Follow-Up of the DANISH Trial. JACC Heart Fail. 2022 Mar;10(3):161-171. doi: 10.1016/j.jchf.2022.01.003. PMID 35241243
- [Derived] Yafasova A, Butt JH, Elming MB, Nielsen JC, Haarbo J, Videbaek L, Olesen LL, Steffensen FH, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Egstrup K, Gustafsson F, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S, Thune JJ, Kober L. Long-Term Follow-Up of DANISH (The Danish Study to Assess the Efficacy of ICDs in Patients With Nonischemic Systolic Heart Failure on Mortality). Circulation. 2022 Feb 8;145(6):427-436. doi: 10.1161/CIRCULATIONAHA.121.056072. Epub 2021 Dec 9. PMID 34882430
- [Derived] Bundgaard JS, Thune JJ, Gislason G, Fosbol EL, Torp-Pedersen C, Aagaard D, Nielsen JC, Haarbo J, Thogersen AM, Videbaek L, Jensen G, Olesen LL, Kristensen SL, Pedersen SS, Kober L, Mogensen UM. Quality of life and the associated risk of all-cause mortality in nonischemic heart failure. Int J Cardiol. 2020 Apr 15;305:92-98. doi: 10.1016/j.ijcard.2020.02.008. Epub 2020 Feb 4. PMID 32046910
- [Derived] Elming MB, Thogersen AM, Videbaek L, Bruun NE, Eiskjaer H, Haarbo J, Egstrup K, Gustafsson F, Hastrup Svendsen J, Hofsten DE, Pehrson S, Nielsen JC, Kober L, Thune JJ. Duration of Heart Failure and Effect of Defibrillator Implantation in Patients With Nonischemic Systolic Heart Failure. Circ Heart Fail. 2019 Sep;12(9):e006022. doi: 10.1161/CIRCHEARTFAILURE.119.006022. Epub 2019 Sep 10. PMID 31500444
- [Derived] Kristensen SL, Levy WC, Shadman R, Nielsen JC, Haarbo J, Videbaek L, Bruun NE, Eiskjaer H, Wiggers H, Brandes A, Thogersen AM, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S, Signorovitch J, Kober L, Thune JJ. Risk Models for Prediction of Implantable Cardioverter-Defibrillator Benefit: Insights From the DANISH Trial. JACC Heart Fail. 2019 Aug;7(8):717-724. doi: 10.1016/j.jchf.2019.03.019. Epub 2019 Jul 10. PMID 31302052
- [Derived] Elming MB, Hammer-Hansen S, Voges I, Nyktari E, Raja AA, Svendsen JH, Pehrson S, Signorovitch J, Kober LV, Prasad SK, Thune JJ. Right Ventricular Dysfunction and the Effect of Defibrillator Implantation in Patients With Nonischemic Systolic Heart Failure. Circ Arrhythm Electrophysiol. 2019 Mar;12(3):e007022. doi: 10.1161/CIRCEP.118.007022. PMID 30866666
- [Derived] Elming MB, Nielsen JC, Haarbo J, Videbaek L, Korup E, Signorovitch J, Olesen LL, Hildebrandt P, Steffensen FH, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Egstrup K, Videbaek R, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S, Kober L, Thune JJ. Age and Outcomes of Primary Prevention Implantable Cardioverter-Defibrillators in Patients With Nonischemic Systolic Heart Failure. Circulation. 2017 Nov 7;136(19):1772-1780. doi: 10.1161/CIRCULATIONAHA.117.028829. Epub 2017 Sep 6. PMID 28877914
- [Derived] Kober L, Thune JJ, Nielsen JC, Haarbo J, Videbaek L, Korup E, Jensen G, Hildebrandt P, Steffensen FH, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Egstrup K, Videbaek R, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S; DANISH Investigators. Defibrillator Implantation in Patients with Nonischemic Systolic Heart Failure. N Engl J Med. 2016 Sep 29;375(13):1221-30. doi: 10.1056/NEJMoa1608029. Epub 2016 Aug 27. PMID 27571011